CLINICAL TRIAL: NCT02828020
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Single Attack Study to Evaluate the Efficacy, Safety, and Tolerability of Oral Ubrogepant in the Acute Treatment of Migraine
Brief Title: Efficacy, Safety, and Tolerability Study of Oral Ubrogepant in the Acute Treatment of Migraine
Acronym: ACHIEVE I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UBR-MD-01
Record Dates: First submitted 2016-07-07; First posted 2016-07-11 (Estimated); Results first posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Migraine, With or Without Aura
MeSH Terms: conditions — Migraine Disorders | interventions — ubrogepant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ubrogepant 50 mg (Experimental): 1 ubrogepant 50 mg tablet and 1 placebo-matching ubrogepant 50 mg tablet, orally for treatment of a qualifying migraine attack. Participants had the option to take a second dose, 2 placebo-matching ubrogepant tablets or rescue medication, orally 2 to 48 hours after initial treatment.
  Interventions: Drug: Ubrogepant; Drug: Placebo-matching Ubrogepant
- Ubrogepant 100 mg (Experimental): 2 Ubrogepant 50 mg tablets, orally for treatment of a qualifying migraine attack. Participants had the option to take a second dose, 2 placebo-matching ubrogepant tablets or rescue medication, orally 2 to 48 hours after initial treatment.
  Interventions: Drug: Ubrogepant; Drug: Placebo-matching Ubrogepant
- Placebo (Placebo Comparator): 2 placebo-matching ubrogepant 50 mg tablets, orally for treatment of a qualifying migraine attack. Participants had the option to take 2-placebo-matching ubrogepant tablets or rescue medication, orally 2 to 48 hours after initial treatment.
  Interventions: Drug: Placebo-matching Ubrogepant

INTERVENTIONS:
Drug: Ubrogepant — 50 mg ubrogepant tablet(s) orally for the treatment of a qualifying migraine attack.
  Arms: Ubrogepant 100 mg; Ubrogepant 50 mg
Drug: Placebo-matching Ubrogepant — Placebo-matching ubrogepant tablet(s) orally for the treatment of a qualifying migraine attack.

SUMMARY:
This study will evaluate the efficacy, safety, and tolerability of 2 doses of ubrogepant (50 and 100 mg) compared to placebo for the acute treatment of a single migraine attack.

ELIGIBILITY:
Inclusion Criteria:

* At least a 1-year history of migraine with or without aura consistent with a diagnosis according to the International Classification of Headache Disorders, 3rd edition, beta version
* Migraine onset before age 50
* History of migraines typically lasting between 4 and 72 hours if untreated or treated unsuccessfully and migraine episodes are separated by at least 48 hours of headache pain freedom
* History of 2 to 8 migraine attacks per month with moderate to severe headache pain in each of the previous 3 months.

Exclusion Criteria:

* Difficulty distinguishing migraine headache from other headaches
* Has taken medication for acute treatment of headache (including acetaminophen, nonsteroidal anti-inflammatory drugs [NSAIDs], triptans, ergotamine, opioids, or combination analgesics) on 10 or more days per month in the previous 3 months
* Has a history of migraine aura with diplopia or impairment of level of consciousness, hemiplegic migraine, or retinal migraine
* Has a current diagnosis of new persistent daily headache, trigeminal autonomic cephalgia (eg, cluster headache), or painful cranial neuropathy
* Required hospital treatment of a migraine attack 3 or more times in the previous 6 months
* Has a chronic non-headache pain condition requiring daily pain medication
* Has a history of malignancy in the prior 5 years, except for adequately treated basal cell or squamous cell skin cancer, or in situ cervical cancer
* Has a history of any prior gastrointestinal conditions (eg, diarrhea syndromes, inflammatory bowel disease) that may affect the absorption or metabolism of investigational product; participants with prior gastric bariatric interventions which have been reversed are not excluded
* Has a history of hepatitis within previous 6 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1672 (Actual)
Dates: Start 2016-07-22 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2017-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adele Thorpe, Study Director — Allergan
Locations (90):
- United States (90):
  - Clinical Research Advantage, Inc./Desert Clinical Research, LLC., Mesa, Arizona
  - Xenoscience, Inc., Phoenix, Arizona
  - Clinical Research Advantage, Inc./Orange Grove Family Practice, Tucson, Arizona
  - Principals Research Group, Inc., Hot Springs, Arkansas
  - KLR Business Group, Inc. dba Arkansas Clinical Research, Little Rock, Arkansas
  - The Research Center of Southern California, LLC, Carlsbad, California
  - Med Center, Carmichael, California
  - T. Joseph Raoof MD, Inc./Encino Research Center, Encino, California
  - Neurology Center of North Orange County, Fullerton, California
  - Behavioral Research Specialists, LLC, Glendale, California
  - Prime Care Clinical Research, Laguna Hills, California
  - Collaborative Neuroscience Network, LLC., Long Beach, California
  - Synergy San Diego, National City, California
  - Newport Beach Clinical Research Associates, Inc., Newport Beach, California
  - North County Clinical Research, Oceanside, California
  - Medical Center for Clinical Research, San Diego, California
  - CA Medical Clinic for Headache, Santa Monica, California
  - Southern California Research LLC, Simi Valley, California
  - Encompass Clinical Research, Spring Valley, California
  - Alpine Clinical Research Center, Inc., Boulder, Colorado
  - Colorado Springs Neurological Associates, Colorado Springs, Colorado
  - Delta Waves, Inc, Colorado Springs, Colorado
  - Denver Neurological Research, Denver, Colorado
  - Associated Neurologists, P.C., Danbury, Connecticut
  - Associated Neurolgists of Southern Connecticut, PC, Fairfield, Connecticut
  - Sarkis Clinical Trials, Gainesville, Florida
  - CPI MD Clinical, Hallandale, Florida
  - Infinity Clinical Research, LLC, Hollywood, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Palm Beach Neurological Center/Advanced Research Consultants, Inc., Palm Beach Gardens, Florida
  - Meridien Research, Spring Hill, Florida
  - University of South Florida, Tampa, Florida
  - Meridien Research, Tampa, Florida
  - Neurology Research Institute, West Palm Beach, Florida
  - Midtown Neurology, Atlanta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Deaconess Clinic, Medical Office Building 1 Research Institute, Newburgh, Indiana
  - Rowe Neurology Institute, Lenexa, Kansas
  - Kansas Institute of Research, Overland Park, Kansas
  - College Park Family Care Center Physicians Group - Neurology Research Department, Overland Park, Kansas
  - Kentucky Pediatric/Adult Research, Bardstown, Kentucky
  - Pharmasite Research, Inc., Baltimore, Maryland
  - Boston Clinical Trials, Boston, Massachusetts
  - Northeast Medical Research Associates, Inc, South Dartmouth, Massachusetts
  - MedVadis Research Corporation, Watertown, Massachusetts
  - Michigan Head-Pain & Neurological Institute, Ann Arbor, Michigan
  - Beyer Research, Kalamazoo, Michigan
  - Clinical Research Institute, Inc., Minneapolis, Minnesota
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - Clinvest Research, LLC, Springfield, Missouri
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Clinical Research Advantage, Inc./Diagnostic Center of Medicine - Durango, Las Vegas, Nevada
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Albuquerque Neuroscience, Inc., Albuquerque, New Mexico
  - Regional Clinical Research, Inc., Endwell, New York
  - Central New York Clinical Research, Manlius, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - Neurology Associates, P.A., Hickory, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - PMG Research of Winston-Salem, LLC., Winston-Salem, North Carolina
  - Neuro-Behavioral Clinical Research, Inc., Canton, Ohio
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Aventiv Research, Inc, Columbus, Ohio
  - Ohio Clinical Research, LLC, Lyndhurst, Ohio
  - MPH IPS Research Company, Oklahoma City, Oklahoma
  - NPC Research, Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Summit Research Network, Portland, Oregon
  - Oregon Center For Clinical Investigations Inc. (OCCI, Inc.), Portland, Oregon
  - Clinical Research of Philadelphia, LLC, Philadelphia, Pennsylvania
  - BTC of Lincoln, Lincoln, Rhode Island
  - WR-ClinSearch, LLC, Chattanooga, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas
  - Tekton Research, Inc., Austin, Texas
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - Red Star Research, LLC, Lake Jackson, Texas
  - Clinical Trials Texas, Inc, San Antonio, Texas
  - Road Runner Research, Ltd., San Antonio, Texas
  - J. Lewis Research, Inc. / Foothill Family Clinic Draper, Draper, Utah
  - Granger Medical Clinic-Riverton, Riverton, Utah
  - Optimum Clinical Research, Inc., Salt Lake City, Utah
  - Highland Clinical Research, Salt Lake City, Utah
  - Tidewater Integrated Medical Research, Virginia Beach, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - The Polyclinic Madison Center, Seattle, Washington

REFERENCES:
- [Derived] Goadsby PJ, Jurgens TP, Brand-Schieber E, Nagy K, Liu Y, Boinpally R, Stodtmann S, Trugman JM. Efficacy of ubrogepant and atogepant in males and females with migraine: A secondary analysis of randomized clinical trials. Cephalalgia. 2025 Feb;45(2):3331024251320610. doi: 10.1177/03331024251320610. PMID 39982105
- [Derived] Johnston KM, Powell L, Popoff E, Harris L, Croop R, Coric V, L'Italien G. Rimegepant, Ubrogepant, and Lasmiditan in the Acute Treatment of Migraine Examining the Benefit-Risk Profile Using Number Needed to Treat/Harm. Clin J Pain. 2022 Nov 1;38(11):680-685. doi: 10.1097/AJP.0000000000001072. PMID 36125279
- [Derived] Lipton RB, Singh RBH, Revicki DA, Zhao S, Shewale AR, Lateiner JE, Dodick DW. Functionality, satisfaction, and global impression of change with ubrogepant for the acute treatment of migraine in triptan insufficient responders: a post hoc analysis of the ACHIEVE I and ACHIEVE II randomized trials. J Headache Pain. 2022 Apr 25;23(1):50. doi: 10.1186/s10194-022-01419-7. PMID 35468729
- [Derived] Blumenfeld AM, Knievel K, Manack Adams A, Severt L, Butler M, Lai H, Dodick DW. Ubrogepant Is Safe and Efficacious in Participants Taking Concomitant Preventive Medication for Migraine: A Pooled Analysis of Phase 3 Trials. Adv Ther. 2022 Jan;39(1):692-705. doi: 10.1007/s12325-021-01923-3. Epub 2021 Dec 7. PMID 34874514
- [Derived] Hutchinson S, Silberstein SD, Blumenfeld AM, Lipton RB, Lu K, Yu SY, Severt L. Safety and efficacy of ubrogepant in participants with major cardiovascular risk factors in two single-attack phase 3 randomized trials: ACHIEVE I and II. Cephalalgia. 2021 Aug;41(9):979-990. doi: 10.1177/03331024211000311. Epub 2021 Apr 19. PMID 33874756
- [Derived] Hutchinson S, Dodick DW, Treppendahl C, Bennett NL, Yu SY, Guo H, Trugman JM. Ubrogepant for the Acute Treatment of Migraine: Pooled Efficacy, Safety, and Tolerability From the ACHIEVE I and ACHIEVE II Phase 3 Randomized Trials. Neurol Ther. 2021 Jun;10(1):235-249. doi: 10.1007/s40120-021-00234-7. Epub 2021 Feb 20. PMID 33608814
- [Derived] Goadsby PJ, Blumenfeld AM, Lipton RB, Dodick DW, Kalidas K, M Adams A, Jakate A, Liu C, Szegedi A, Trugman JM. Time course of efficacy of ubrogepant for the acute treatment of migraine: Clinical implications. Cephalalgia. 2021 Apr;41(5):546-560. doi: 10.1177/0333102420970523. Epub 2020 Nov 26. PMID 33241721
- [Derived] Dodick DW, Lipton RB, Ailani J, Lu K, Finnegan M, Trugman JM, Szegedi A. Ubrogepant for the Treatment of Migraine. N Engl J Med. 2019 Dec 5;381(23):2230-2241. doi: 10.1056/NEJMoa1813049. PMID 31800988
- See also: More Information — http://www.allerganclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period
Arm/Group | Placebo | Ubrogepant 50 mg | Ubrogepant 100 mg
Started | 559 | 556 | 557
Safety Population: Received Study Drug | 485 | 466 | 485
Completed | 479 | 457 | 479
Not Completed | 80 | 99 | 78
Not completed — Adverse Event | 3 | 1 | 1
Not completed — Withdrawal of Consent | 10 | 14 | 9
Not completed — Lost to Follow-up | 21 | 24 | 18
Not completed — Lack of Qualifying Event | 44 | 53 | 43
Not completed — Pregnancy | 0 | 2 | 0
Not completed — Protocol Violation | 2 | 4 | 7
Not completed — Other Miscellaneous Reasons | 0 | 1 | 0
Period: Safety Follow-up Period
Arm/Group | Placebo | Ubrogepant 50 mg | Ubrogepant 100 mg
Started | 480 (1 participant who did not complete the Treatment Period, was counted in the Safety Follow-up Period.) | 458 (1 participant who did not complete the Treatment Period, was counted in the Safety Follow-up Period.) | 480 (1 participant who did not complete the Treatment Period, was counted in the Safety Follow-up Period.)
Completed | 460 | 440 | 461
Not Completed | 20 | 18 | 19
Not completed — Withdrawal of Consent | 10 | 8 | 7
Not completed — Lost to Follow-up | 9 | 8 | 11
Not completed — Protocol Violation | 0 | 2 | 1
Not completed — Other Miscellaneous Reasons | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ubrogepant 50 mg | Ubrogepant 100 mg | Total
Number analyzed (Participants) | 559 | 556 | 557 | 1672
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (11.9) | 40.2 (12.0) | 40.7 (12.4) | 40.7 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 491 | 493 | 479 | 1463
  Male | 68 | 63 | 78 | 209
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 471 | 459 | 447 | 1377
  Black or African American | 65 | 77 | 88 | 230
  Asian | 10 | 9 | 8 | 27
  American Indian or Alaska Native | 3 | 3 | 5 | 11
  Native Hawaiian/Other Pacific Islander | 3 | 1 | 5 | 9
  Multiple | 7 | 7 | 4 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 60 | 67 | 66 | 193
  Not Hispanic or Latino | 499 | 489 | 491 | 1479

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Pain Freedom at 2 Hours After Initial Dose
Description: Pain freedom was defined as a reduction in headache severity from moderate/severe at baseline to no pain at 2 hours after the initial dose. Participants were provided with an electronic diary (eDiary) to rate headache severity on a scale from no pain to severe pain. Number analyzed is the number of participants with non-missing postdose pain severity assessment at or before 2 hours after initial dose.
Time Frame: Baseline (Predose) to 2 hours after initial dose
Population: Modified Intent-to-Treat (mITT) population included all randomized participants who received at least 1 dose of study drug, recorded a baseline migraine headache severity measurement, and had ≥ 1 postdose migraine headache severity or migraine-associated symptom measurement at or before the 2-hour timepoint, last observation carried forward (LOCF).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ubrogepant 50 mg | Ubrogepant 100 mg
Number analyzed (Participants) | 456 | 422 | 448
percentage of participants | 11.8 | 19.2 | 21.2
Statistical Analysis 1: Comparison: Placebo vs Ubrogepant 50 mg; Test type: Superiority; p = 0.0023, Regression, Logistic — P-value was adjusted for multiple comparisons across primary and secondary endpoints and multiple doses; Treatment group, historical triptan response, medication use for migraine prevention, baseline headache severity were explanatory variables in model; Odds Ratio (OR) = 1.83, 95% CI 2-sided [1.25 to 2.66]
Statistical Analysis 2: Comparison: Placebo vs Ubrogepant 100 mg; Test type: Superiority; p = 0.0003, Regression, Logistic — P-value was adjusted for multiple comparisons across primary and secondary endpoints and multiple doses; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.04, 95% CI 2-sided [1.41 to 2.95]

2. Primary Outcome: Percentage of Participants With Absence of the Most Bothersome Migraine-Associated Symptom Identified at Baseline at 2-Hours After Initial Dose
Description: The most bothersome migraine-associated symptom was the symptom (photophobia, phonophobia or nausea) present at pre-dose baseline identified by the participant to be 'most bothersome'. Participants were provided with an eDiary to record absence or presence of migraine-associated symptoms. Number analyzed is the number of participants with non-missing postdose most bothersome migraine-associated symptoms.
Time Frame: Baseline (Predose) to 2 hours after initial dose
Population: mITT population included all randomized participants who received at least 1 dose of investigational product, recorded a baseline migraine headache severity measurement, and had ≥ 1 postdose migraine headache severity or migraine-associated symptom measurement at or before the 2-hour timepoint, LOCF.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ubrogepant 50 mg | Ubrogepant 100 mg
Number analyzed (Participants) | 454 | 420 | 448
percentage of participants | 27.8 | 38.6 | 37.7
Statistical Analysis 1: Comparison: Placebo vs Ubrogepant 50 mg; Test type: Superiority; p = 0.0023, Regression, Logistic — P-value was adjusted for multiple comparisons across primary and secondary endpoints and multiple doses; Treatment group, historical triptan response, migraine prevention medication, baseline headache severity, underlying symptom as explanatory variables; Odds Ratio (OR) = 1.70, 95% CI 2-sided [1.27 to 2.28]
Statistical Analysis 2: Comparison: Placebo vs Ubrogepant 100 mg; Test type: Superiority; p = 0.0023, Regression, Logistic — P-value was adjusted for multiple comparisons across primary and secondary endpoints and multiple doses; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.63, 95% CI 2-sided [1.22 to 2.17]

3. Secondary Outcome: Percentage of Participants With Pain Relief at 2 Hours After the Initial Dose
Description: Pain relief was defined as a reduction of a moderate/severe migraine headache to a mild headache or to no headache. Participants were provided with an eDiary to rate headache severity on a scale from no pain to severe pain. Number analyzed is the number of participants with non-missing pain severity assessment at or before 2 hours after initial dose.
Time Frame: Baseline (Predose) to 2 hours after initial dose
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ubrogepant 50 mg | Ubrogepant 100 mg
Number analyzed (Participants) | 456 | 422 | 448
percentage of participants | 49.1 | 60.7 | 61.4
Statistical Analysis 1: Comparison: Placebo vs Ubrogepant 50 mg; Test type: Superiority; p = 0.0023, Regression, Logistic — P-value was adjusted for multiple comparisons across primary and secondary endpoints and multiple doses; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.69, 95% CI 2-sided [1.28 to 2.23]
Statistical Analysis 2: Comparison: Placebo vs Ubrogepant 100 mg; Test type: Superiority; p = 0.0023, Regression, Logistic — P-value was adjusted for multiple comparisons across primary and secondary endpoints and multiple doses; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.69, 95% CI 2-sided [1.28 to 2.21]

4. Secondary Outcome: Percentage of Participants With Sustained Pain Relief From 2 to 24 Hours After Initial Dose
Description: Sustained pain relief was defined as a pain relief at 2 hours with no administration of either rescue medication or the second dose of study drug, and with no occurrence thereafter of a moderate/severe headache up to 24 hours after dosing with study drug. Participants were provided with an eDiary to rate headache severity on a scale from no pain to severe pain. Determinable cases: participants for whom sustained pain relief from 2 to 24 hours status can be determined based on the observed headache severity at scheduled time points, use of rescue medication or optional second dose between 2 and 24 hours, and the answer to the headache recurrence question at 24 hours. Number analyzed is the number of participants with determinable sustained pain relief from 2 to 24 hours after initial dose.
Time Frame: 2 to 24 hours after initial dose
Population: mITT population included all randomized participants who received at least 1 dose of investigational product, recorded a baseline migraine headache severity measurement, and had ≥ 1 postdose migraine headache severity or migraine-associated symptom measurement at or before the 2-hour timepoint, determinable cases.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ubrogepant 50 mg | Ubrogepant 100 mg
Number analyzed (Participants) | 447 | 413 | 434
percentage of participants | 20.8 | 36.3 | 38.0
Statistical Analysis 1: Comparison: Placebo vs Ubrogepant 50 mg; Test type: Superiority; p = 0.0023, Regression, Logistic — P-value was adjusted for multiple comparisons across primary and secondary endpoints and multiple doses; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.25, 95% CI 2-sided [1.65 to 3.07]
Statistical Analysis 2: Comparison: Placebo vs Ubrogepant 100 mg; Test type: Superiority; p = 0.0023, Regression, Logistic — P-value was adjusted for multiple comparisons across primary and secondary endpoints and multiple doses; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.39, 95% CI 2-sided [1.77 to 3.24]

5. Secondary Outcome: Percentage of Participants With Sustained Pain Freedom From 2 to 24 Hours After Initial Dose
Description: Sustained pain freedom was defined as a pain freedom at 2 hours with no administration of either rescue medication or the second dose of study drug, and with no occurrence thereafter of a mild/moderate/severe headache up to 24 hours after dosing with study drug. Participants were provided with an eDiary to rate headache severity on a scale from no pain to severe pain. Determinable cases: participants for whom sustained pain relief from 2 to 24 hours status can be determined based on the observed headache severity at scheduled time points, use of rescue medication or optional second dose between 2 and 24 hours, and the answer to the headache recurrence question at 24 hours. Number analyzed is the number of participants with determinable sustained pain freedom from 2 to 24 hours after initial dose.
Time Frame: 2 to 24 hours after initial dose
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ubrogepant 50 mg | Ubrogepant 100 mg
Number analyzed (Participants) | 452 | 418 | 441
percentage of participants | 8.6 | 12.7 | 15.4
Statistical Analysis 1: Comparison: Placebo vs Ubrogepant 50 mg; Test type: Superiority; p = 0.0577, Regression, Logistic — P-value was adjusted for multiple comparisons across primary and secondary endpoints and multiple doses; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.57, 95% CI 2-sided [1.01 to 2.44]
Statistical Analysis 2: Comparison: Placebo vs Ubrogepant 100 mg; Test type: Superiority; p = 0.0037, Regression, Logistic — P-value was adjusted for multiple comparisons across primary and secondary endpoints and multiple doses; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.95, 95% CI 2-sided [1.28 to 2.97]

6. Secondary Outcome: Percentage of Participants With the Absence of Photophobia at 2 Hours After the Initial Dose
Description: Photophobia was defined as sensitivity to light, a migraine-associated symptom. Participants were provided with an eDiary to record absence or presence photophobia. Number analyzed is the number of participants with non-missing postdose photophobia assessment at or before 2 hours after initial dose.
Time Frame: 2 hours after initial dose
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ubrogepant 50 mg | Ubrogepant 100 mg
Number analyzed (Participants) | 456 | 423 | 448
percentage of participants | 31.4 | 40.7 | 45.8
Statistical Analysis 1: Comparison: Placebo vs Ubrogepant 50 mg; Test type: Superiority; p = 0.0577, Regression, Logistic — P-value was adjusted for multiple comparisons across primary and secondary endpoints and multiple doses; Treatment group, historical triptan response, migraine prevention medication, baseline headache severity, photophobia were explanatory variables; Odds Ratio (OR) = 1.63, 95% CI 2-sided [1.22 to 2.19]
Statistical Analysis 2: Comparison: Placebo vs Ubrogepant 100 mg; Test type: Superiority; p = 0.0037, Regression, Logistic — P-value was adjusted for multiple comparisons across primary and secondary endpoints and multiple doses; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 1.81, 95% CI 2-sided [1.36 to 2.42]

7. Secondary Outcome: Percentage of Participants With the Absence of Phonophobia at 2 Hours After the Initial Dose
Description: Phonophobia was defined as sensitivity to sound, a migraine-associated symptom. Participants were provided with an eDiary to record absence or presence of phonophobia. Number analyzed is the number of participants with non-missing postdose phonophobia assessment at or before 2 hours after initial dose.
Time Frame: 2 hours after initial dose
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ubrogepant 50 mg | Ubrogepant 100 mg
Number analyzed (Participants) | 456 | 423 | 448
percentage of participants | 47.1 | 57.9 | 54.5
Statistical Analysis 1: Comparison: Placebo vs Ubrogepant 50 mg; Test type: Superiority; p = 0.0577, Regression, Logistic — P-value was adjusted for multiple comparisons across primary and secondary endpoints and multiple doses; Treatment group, historical triptan response, migraine prevention medication, baseline headache severity, phonophobia were explanatory variables; Odds Ratio (OR) = 1.56, 95% CI 2-sided [1.16 to 2.09]
Statistical Analysis 2: Comparison: Placebo vs Ubrogepant 100 mg; Test type: Superiority; p = 0.0577, Regression, Logistic — P-value was adjusted for multiple comparisons across primary and secondary endpoints and multiple doses; [statistical method as in outcome 7, analysis 1]; Odds Ratio (OR) = 1.47, 95% CI 2-sided [1.10 to 1.95]

8. Secondary Outcome: Percentage of Participants With Absence of Nausea at 2 Hours After the Initial Dose
Description: Nausea was a migraine-associated symptom. Participants were provided with an eDiary to record absence or presence of nausea. Number analyzed is the number of participants with non-missing postdose nausea assessment at or before 2 hours after initial dose.
Time Frame: 2 hours after initial dose
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ubrogepant 50 mg | Ubrogepant 100 mg
Number analyzed (Participants) | 456 | 423 | 448
percentage of participants | 62.3 | 70.2 | 69.2
Statistical Analysis 1: Comparison: Placebo vs Ubrogepant 50 mg; Test type: Superiority; p = 0.0962, Regression, Logistic — P-value was adjusted for multiple comparisons across primary and secondary endpoints and multiple doses; Treatment group, historical triptan response, migraine prevention medication, baseline headache severity, nausea were explanatory variables; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.96 to 1.79]
Statistical Analysis 2: Comparison: Placebo vs Ubrogepant 100 mg; Test type: Superiority; p = 0.0962, Regression, Logistic — P-value was adjusted for multiple comparisons across primary and secondary endpoints and multiple doses; [statistical method as in outcome 8, analysis 1]; Odds Ratio (OR) = 1.35, 95% CI 2-sided [1.00 to 1.83]

ADVERSE EVENTS:
Time Frame: From first dose through 30 days after the last dose of study drug (approximately 30 days)
Description: Safety population, all participants who received at least 1 dose of investigational product was used to determine the number of participants at risk for Serious Adverse Events and Other Adverse Events
Arm/Group | Placebo | Ubrogepant 50 mg | Ubrogepant 100 mg
All-Cause Mortality (participants affected / at risk) | 0/485 | 0/466 | 0/485
Serious Adverse Events (participants affected / at risk) | 0/485 | 3/466 | 2/485
Other Adverse Events (participants affected / at risk) | 0/485 | 0/466 | 0/485
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=485) | Ubrogepant 50 mg (N=466) | Ubrogepant 100 mg (N=485)
Appendicitis (Infections and infestations) | 0 | 1 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-05-19): https://cdn.clinicaltrials.gov/large-docs/20/NCT02828020/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-22): https://cdn.clinicaltrials.gov/large-docs/20/NCT02828020/SAP_001.pdf